CLINICAL TRIAL: NCT02096978
Title: A Randomized Controlled Clinical Study Comparing Implant Stability Using Osteotome vs. Conventional Drilling Techniques by Resonance Frequency Analysis
Brief Title: Comparing Implant Stability Using Two Accepted Techniques for Implant Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120100304
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Implant
Keywords: Implant; Stability; placement; Osteotome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteotome preparation (Experimental): Procedure/Surgery: Preparing the osteotomy to accept a standard implant device
  Interventions: Procedure: Preparing the osteotomy to accept a standard implant device
- Drill preparation (Active Comparator): Preparing the osteotomy to accept a standard implant device
  Interventions: Procedure: Preparing the osteotomy to accept a standard implant device

INTERVENTIONS:
Procedure: Preparing the osteotomy to accept a standard implant device — Preparing the osteotomy with one of two randomly assigned protocols

SUMMARY:
The study will be conducted to compare two alternative techniques for dental implant placement. Both of the techniques - Osteotome and Conventional Drilling Techniques for the preparation of the implant sites (osteotomies) are accepted standards of care. The goal of the study will be to compare implant stabilities achieved with two techniques by measuring resonance frequency for each implant placed using the diagnostic device, the Osstell machine, that measures "stiffness" of the bone/implant system non-invasively. The data are represented in a quantitative value - implant stability quotient (ISQ), where a higher value indicated a higher implant stability. Since it has been well documented in the scientific literature that primary (at the time of implant placement) implant stability is a strong prerequisite for implant success (osseointegration and subsequent function on loading), the results of this study will guide the implant team in choosing the right surgical treatment protocol - the protocol that will be aimed for higher implant stability, and, therefore, for higher long-term implant success.

DETAILED DESCRIPTION:
With the emergence of one stage surgical approach to implant placements with immediate loading (IL), the importance of achieving uncompromised primary stability, especially in poor bone density (D3, D4), cannot be underestimated. Degidi et al. showed that poor quality bone was related to increased marginal bone loss and inferior clinical outcomes for IL implants. In a 5 year retrospective study, Elkhoury et al. found that one of the significant clinical parameters, associated with success of plasma-sprayed cylindrical dental implants was higher bone density (P<0.0001). Hermann et al evaluated 487 implants randomly selected from a research created database that used different implant placements protocols placed over a 5 year period and found out that implant failures were primarily associated with negative bone-related patient factors: jawbone quality and shape.

Two bone types that fall in the negative bone-related factors are types D3 and D4. D3 type bone, which consists of thin porous cortical and fine trabecular bone, according to the Misch bone density classification, is most prevalent in anterior maxilla and posterior regions of maxilla and mandible. In a review of 73 published articles, by Esposito et al., biological factors that contribute to failures of osseointegrated oral implants, the authors confirmed that maxillas, due to their poor bone density, have almost 3 times more implant failures than mandibles.

In planning the case, it is very important to differentiate between bone quality and bone density. Bone quality comprises bone metabolism, cell turn over, mineralization, maturation, intercellular matrix, and vascularization and while all of these factors influence implant success, it is valuable to be able to isolate them in order to be able to investigate their individual contributions to implant outcomes.

The development of three-dimensional imaging, such as Computed Tomography (CT) and Cone Beam Computed Tomography (CBCT) has recently became the standard of care during pre-surgical phase, at implant planning stage. It enables an implant team to provide the most precise and reliable diagnostic information on the patient's vital anatomy, bone quality and bone quantity at the proposed implant sites. In 95% of cases that use CT, bone quantity determination is to +/- 1 mm of accuracy, compared to only 30% of cases that use panoramic radiology.

A comprehensive review of 45 manuscripts by Molly that investigated and discussed the relationship between bone density and primary implant stability concluded that there is a significant correlation exists between bone density, primary stability, and implant outcomes.

One of the necessary, although not sufficient, determinants of implant success is successful osseointegration, which was defined by Albrektsson as a "direct functional and structural connection between living bone and the surface of a load-bearing implant". However, non-invasive determination of the degree of osseointegration is not yet possible in clinical practice. Therefore, assessments of primary and secondary implant stability could indirectly provide clinicians with the degree of future and present osseointegration, respectively.

Stability of an implant can be defined as "its capacity to withstand loading forces in axial, lateral, and rotational directions". It can be subdivided into "primary" and "secondary". Primary stability has been coined by Branemark as a prerequisite to achieve osseointegration (Branemark et al. 1977). It is the stability of an implant body that is achieved during implant installation by the physical congruence between the surgically created bone bed (osteotomy) and the implant, which depends on surgical technique, bone density, and macroscopic implant design. It also can serve as a predictor of future osseointegration. Secondary implant stability is the stability that is gradually achieved after osseointegration of an implant, and is highly correlated with bone to implant contact surface area, depending on microscopic implant design since the bone is being formed inside implants threads.

In order to provide objective measurements of primary or second implant stabilities, resonance-frequency analysis (RFA) has been introduced. In addition to providing quantitative information about the degree of primary implant stability, it is also useful to monitor implant osseointegration during the healing phase in order to help establish individual loading time protocols. Nedir et al., evaluated predictability of osseointegration as measured by RFA, which quantitates the implant stability, and the authors suggested that implants with ISQ>49 should osseointegrate predictably, when left submerged to heal for 3 months, and implants with ISQ>54 might be immediately loaded. Rodrigo et al., used clinical evaluation and RFA measurements to diagnose implant stability and its impact on implant survival and concluded that only secondary stability RFA values were good predictors of implant outcomes.

One of the classical surgical protocols in the posterior maxilla is the osteotome technique that was introduced by Summers in 1997 in order to be able to take advantage of the poor bone quality by relocating the available bone to accommodate the needs of the surgical procedure. Since the implants were placed without drilling, it was meant to be an essentially "heatless" procedure that compacted the bone adjacent to the prepared osteotomy, thus, improving "osseointegration". Since then, the procedure has become successfully established as a surgical routine, but it has mostly been used in cases where either ridge expansion, or internal sinus elevation is needed. It is crucial to point out that only divergent osteotomes will be able to compact the bone laterally without crushing the bone and that since the technique in itself provides bone compaction immediately adjacent to the implant site, it might be beneficial to utilize osteotomes in implant protocols even when sinus elevation or ridge augmentation are not necessary.

Pjetursson et al. utilized osteotome technique and in their study more than 90% of patients were satisfied with the treatment and reported that they would undergo the same procedure again and recommend it to their family members or friends, thus, demonstrating that osteotome technique has perfect patient acceptance.

In the present human case control study the investigators will compare the ISQ values of maxillary implants placed using the osteotome technique, described by Drew et al. and conventional drilling techniques. Our hypothesis is that due to the divergent design of the osteotomes, bone quality will be improved, therefore, improving bone-to-implant contact ratio, which will be illustrated by higher ISQ values in the osteotome group.

Hypotheses:

1. Primary implant stability, measured by resonance frequency analysis (RFA) at the time of implant placement is higher in the implants placed with the osteotomes (O Group) vs. conventional drilling (D group) (ISQprimary (O) > ISQprimary (D)).
2. Secondary implant stability, measured by resonance frequency analysis (RFA) at 30, 60, and 90 days, is higher in the implants placed with the osteotomes vs. conventional drilling (ISQsecondary (O) > ISQsecondary (D)).

Patients will have 1 implant fixtures Biomet 3 I Osseotite Certain Prevail (same diameter and length: 4x10 mm) placed in the maxilla (upper jaw) by randomly assigned two experienced surgeons. Randomization will be done so that the surgeon will place implants in randomly assigned patients (half implants using Osteotome technique and half implants using Drilling technique). Fixtures will be randomly assigned to either Osteotome (O) or Conventional Drilling (D) group using a randomization plan developed online from www.randomization.com. Healing abutments (2 mm supragingivally) will be placed if the primary stability will be attained.

In cases, RFA measurement is less than 49 ISQ, the implants will be submerged and the second measurement will be done after implant uncovery at 90 days. All subjects will have completed Phase I therapy (non-surgical) with no active periodontal disease and/or caries.

A diagnostic wax up will be made for each case and a clear radiographic/surgical template fabricated for three-dimensional analysis and implant placement surgery.

Cone Beam CT scans (ICATvision® software and ICAT Next Generation® machine, Hatfield, PA) as an accepted standard of care, will be done prior to surgery to plan the surgery and to confirm the bone density of type D3 or type D 4 (D 1 and D 2 will be excluded from the study) in Hounsfield units (H.U.). The accepted bone density values and their corresponding bone quality when a medical CT scanning is used are as follows.

D 1 Bone (> 1250 H.U.) D 2 Bone (850-1250 H.U.) D 3 Bone (350-850 H.U.) D 4 Bone (< 400 H.U.) The imaging will verify that adequate horizontal and vertical dimensions of bone are present, prior to surgery. A minimum of 7mm of horizontal bone and a minimum of 12 mm of vertical height will be needed to accommodate a 4x10mm fixture.

Local Anesthesia of 2% Lidocaine with 1:100000epi or 3% Carbocaine without vasoconstrictor buccal and palatal infiltration. Mid-crestal, intra-sulcular incisions extending to one tooth mesial and distal to the surgery site. Full thickness flap reflection. Osteotome group fixtures (O) will be placed according to the technique described by Drew et al. Conventional drilling technique Fixtures will be placed according Biomet 3 I surgical protocol. Final insertion torque of each implant will be recorded in 20, 32, or 45 Ncm by the Biomet 3 I machine, which is utilized for perforation of bone and implant placement. It can only apply finite amount of torque in order to avoid damage to the alveolar bone due to overheating. Healing caps 2 mm supragingivally placed and ISQ values recorded using Osstell device. (If ISQ < 49, the implants will be submerged, and left to osseointegrate for 90 days. Only 0 and 90 days recording will be made). 4-0 Vicryl suture will be used to obtain primary closure.

All fixtures will be placed at 20, 32, or 45 Ncm torque. ISQ values will be recorded by Osstell device at the time of implant placement (0) and at 30. 60, and 90 days. Each ISQ measurement will be repeated twice with two different transducers and the mean ISQ value will be used for the analysis. The transducer will be screwed manually and the measurement device will be directed perpendicularly to the direction of the fixture.

Clinical parameters that will be recorded at 0, 30, 60, and 90 days:

A. Resonance frequency measurements of each implant. B. Final torque Measurements of each implant in Ncm. Soft tissue height (mesio-buccal (MB), buccal(B), disto-buccal(DB), mesio-palatal(MP), palatal(P), disto-palatal (DP)) (measured from the gingival margin to the depth of the pocket). Soft tissue levels measured at MB, B, DB, P, (measured from the soft tissue margin to the mark on the occlusal stent) at 0 and 90 days only. Crestal bone area (bitewing conventional radiography with customized intraoral X ray film holders) All cases will be done with antibiotic premedication (Amoxicillin 2000mg or Zithromax 500mg, 1 hour prior to surgery). Post-op instructions will include Chlorhexidine gluconate 0.15% mouthwash BID for 21 days, pain control medication and an antibiotic. Patients that will develop complications (infection, loss of implant etc…) will be followed up and treated in accordance to the established standard of care.

In the event of mobility the implant will be removed and the site grafted, and implant replaced in 3-6 months at no charge to patient.

Data Analysis:

Data will be analyzed using Two-sample T-test.

ELIGIBILITY:
Inclusion Criteria:

* One maxillary implant fixture per patient indicated by the treatment plan.
* No previous implant attempted in the area
* No previous GBR or sinus lift done
* No GBR or sinus lift needed
* A minimum of 7mm of horizontal bone and a minimum of 12mm of vertical height will be needed to accommodate a 4x10mm fixture.

Exclusion Criteria:

* History of diabetes, HIV+, radiation therapy, smoking, oral/intravenous bisphosphonates intake.
* Pregnant women
* Maxillary bone density of Type D1/Type D2, as determined by a preoperative three-dimensional imaging.
* No grafted sites.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Necessary stability to insert prosthesis by RFA units | 90 days
  Stability to be measured by RFA units

CONTACTS AND LOCATIONS:
Overall Officials: Howard J Drew, DMD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

REFERENCES:
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- [Background] Buchter A, Kleinheinz J, Wiesmann HP, Kersken J, Nienkemper M, Weyhrother Hv, Joos U, Meyer U. Biological and biomechanical evaluation of bone remodelling and implant stability after using an osteotome technique. Clin Oral Implants Res. 2005 Feb;16(1):1-8. doi: 10.1111/j.1600-0501.2004.01081.x. PMID 15642025
- [Background] Stavropoulos A, Nyengaard JR, Lang NP, Karring T. Immediate loading of single SLA implants: drilling vs. osteotomes for the preparation of the implant site. Clin Oral Implants Res. 2008 Jan;19(1):55-65. doi: 10.1111/j.1600-0501.2007.01422.x. Epub 2007 Oct 22. PMID 17956566
- [Background] Devlin H, Horner K, Ledgerton D. A comparison of maxillary and mandibular bone mineral densities. J Prosthet Dent. 1998 Mar;79(3):323-7. doi: 10.1016/s0022-3913(98)70245-8. PMID 9553887